CLINICAL TRIAL: NCT05873907
Title: A Randomized, Double-blind, Placebo-controlled, Single-ascending Dose Study to Evaluate the Safety, Tolerability, Immunogenicity, Pharmacokinetics, and Pharmacodynamics of AMG 592 in Healthy Subjects
Brief Title: A Study to Evaluate the Safety, Tolerability, Immunogenicity, Pharmacokinetics, and Pharmacodynamics of AMG 592 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 20140324
Record Dates: First submitted 2023-05-16; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Chronic Graft-versus-host Disease (cGVHD)
Keywords: Chronic Graft-versus-Host Disease; AMG 592; Inflammatory Conditions
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- AMG 592: Dose 1 (Experimental): Administered as a single dose subcutaneous (SC) injection.
  Interventions: Drug: AMG 592
- AMG 592: Dose 2 (Experimental): Administered as a single dose SC injection.
  Interventions: Drug: AMG 592
- AMG 592: Dose 3 (Experimental): Administered as a single dose SC injection.
  Interventions: Drug: AMG 592
- AMG 592: Dose 4 (Experimental): Administered as a single dose SC injection.
  Interventions: Drug: AMG 592
- AMG 592: Dose 5 (Experimental): Administered as a single dose SC injection.
  Interventions: Drug: AMG 592
- AMG 592: Dose 6 (Experimental): Administered as a single dose SC injection.
  Interventions: Drug: AMG 592
- AMG 592: Dose 7 (Experimental): Administered as a single dose SC injection.
  Interventions: Drug: AMG 592
- AMG 592: Dose 8 (Experimental): Administered as a single dose SC injection.
  Interventions: Drug: AMG 592
- Placebo (Placebo Comparator): Administered as SC injection.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AMG 592 — Administered as SC injection
  Arms: AMG 592: Dose 1; AMG 592: Dose 2; AMG 592: Dose 3; AMG 592: Dose 4; AMG 592: Dose 5; AMG 592: Dose 6; AMG 592: Dose 7; AMG 592: Dose 8
Other: Placebo — Administered as SC injection
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the safety, tolerability and immunogenicity profile of single and multiple dose administrations of AMG 592 in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Males must agree to practice an acceptable method of effective birth control while on study through 2 weeks after receiving the dose of study drug.
* Males must be willing to abstain from sperm donation while on study through 2 weeks after receiving the (last [multiple dose studies]) dose of study drug.
* Male and female subjects ≥ 18 and ≤ 55 years of age with a body mass index (BMI) of ≥ 18.0 and ≤ 32.0 kg/m^2 at the time of screening.
* Females must be of non-reproductive potential (ie, postmenopausal - age ≥ 55 years with cessation of menses for 12 months or more, or according to the definition of "postmenopausal range" for the laboratory involved OR history of hysterectomy; OR history of bilateral oophorectomy).

Exclusion Criteria:

* Positive Hepatitis B Surface Antigen (HepBsAg) (indicative of chronic Hepatitis B) or detectable Hepatitis C virus Ribonucleic acid (RNA) by Polymerase Chain Reaction (PCR) (indicative of active Hepatitis C - screening is generally done by Hepatitis C Antibody (HepCAb), followed by Hepatitis C virus RNA by PCR if HepCAb is positive).
* Positive results for Human Immunodeficiency Virus (HIV).
* Participant has a history of residential exposure to tuberculosis without a documented history of prophylactic treatment of tuberculosis or participant has a positive purified protein derivative (PPD) or QuantiFERON or T-Spot test at Screening. Participants with a documented negative PPD or QuantiFERON or T-Spot test within 4 weeks prior to screening who have no known tuberculosis exposure and have not traveled to an area with tuberculosis do not need to have a test performed at screening.
* Currently receiving treatment in another investigational device or drug study, or less than 30 days or less than 5 half-lives, whichever is longer, since ending treatment on another investigational device or drug study.
* Malignancy except non-melanoma skin cancers, cervical or breast ductal carcinoma in situ within the last 5 years.
* Any active infection for which systemic anti-infectives were used within 4 weeks prior to Day 1.
* Females who are lactating/breastfeeding or who plan to breastfeed while on study through 2 weeks after receiving the dose of study drug.
* Female participants with a positive pregnancy test.
* Males with partners who are pregnant or planning to become pregnant while the participant is on study through 2 weeks after receiving the dose of study drug.
* Has any significant abnormality during the screening physical examination, electrocardiogram (ECG), or laboratory evaluation that in the opinion of the Investigator, in consultation with the Amgen Medical Monitor, would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion.
* Unwilling or unable to abstain from alcohol consumption within 48 hours prior to each visit (including Screening).
* Is a current smoker, has used any nicotine or tobacco containing products (including but not limited to: snuff, chewing tobacco, cigars, cigarettes, pipes, or nicotine patches) within the last 6 months from Screening, and cumulative smoking history is ≥ 10 pack years.
* Unwilling or unable to refrain from strenuous exercise (eg, heavy lifting, weight training, and aerobics) for 72 hours prior to each visit that includes blood collection.
* Has donated or lost ≥ 500 mL of blood or plasma within 8 weeks of administration of the first dose of IP.
* Participants with a known history of autoimmune disease.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2015-10-19 (Actual); Primary Completion 2017-06-16 (Actual); Study Completion 2017-07-28 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events (TEAEs) | Day 1 up to Day 57
  Any clinically significant changes in physical examinations, clinical laboratory tests and vital signs will be recorded as TEAEs.
Number of Participants with Anti-AMG 592 Antibodies | Day 1 up to Day 57
Fold Change from Baseline in Absolute Cell Counts of Regulatory T Cells (Tregs) | One week after AMG 592 administration (up to 7 days)
Fold Change from Baseline in Absolute Cell Counts of Conventional T Cells (Tcons) | One week after AMG 592 administration (up to 7 days)
Fold Change from Baseline in Absolute Cell Counts of Natural Killer Cells (NKs) | One week after AMG 592 administration (up to 7 days)

SECONDARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) of AMG 592 | Day 1 up to Day 57
Time of Maximum Observed Concentration (tmax) of AMG 592 | Day 1 up to Day 57
Area Under the Concentration-time Curve (AUC) of AMG 592 | Day 1 up to Day 57

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- Research Site, Aventura, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com